CLINICAL TRIAL: NCT03018262
Title: Detailed Evaluation of the Neurophysiology of Surround Inhibition in the Human Motor Cortex
Brief Title: Neurophysiology of Surround Inhibition in the Human Motor Cortex
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170031; 17-N-0031
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Normal Physiology
Keywords: Surround Inhibition; Motor Control; Transcranial Magnetic Stimulation (TMS); TMS-Evoked Potential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Healthy Volunteers - Sub-study 1: Healthy Volunteers
  Interventions: Device: TMS - sub-study 1
- Healthy Volunteers - Sub-study 2: Healthy Volunteers
  Interventions: Device: TMS - sub-study 2
- Healthy Volunteers - Sub-study 3: Healthy Volunteers
  Interventions: Device: TMS - sub-study 3

INTERVENTIONS:
Device: TMS - sub-study 1 — TMS pulses will be applied to the motor hotspot of the surround muscle to identify the TMS-evoked potentials corresponding to motor surround inhibition (SI)
  Groups: Healthy Volunteers - Sub-study 1
Device: TMS - sub-study 2 — TMS will be used to stimulate the motor cortex and an inhibitory region of the inferior parietal lobe
  Groups: Healthy Volunteers - Sub-study 2
Device: TMS - sub-study 3 — TMS pulses will be delivered to the primary motor cortex at rest, at the onset of the motor task, or during the motor task
  Groups: Healthy Volunteers - Sub-study 3

SUMMARY:
Background:

Movement disorders have many different causes and symptoms. Researchers still do not fully understand which parts of the brain are involved in fine movement. They want to learn about which brain regions could be abnormal in people with movement disorders.

Objective:

To better understand how the brain controls movement.

Eligibility:

Healthy, right-handed adults age 18-70 years old.

Design:

Participants will be screened with a physical exam and questions about their handedness. They may have a urine test.

Participants will have 1 or 2 clinic visits. The first visit will last about 1.5 hours. The second will last about 3 hours.

Participants will have structural magnetic resonance imaging (MRI). A strong magnetic field and radio waves take pictures of the brain. Participants will lie on a table that slides in and out of a metal cylinder.

Participants may have transcranial magnetic stimulation. A wire coil is held on the scalp. A brief electrical current is passed through the coil and creates a magnetic pulse that stimulates the brain. Participants will wear a pair of glasses or a headband with small sensors so researchers can track head position.

Participants will perform a simple index finger movement task.

Participants may have surface electromyography from at least two hand muscles. Small metal disk or adhesive pad electrodes will be taped to the skin. Participants will be seated in a comfortable chair with their hands placed on a pillow.

Participants may have an electroencephalography. A cap with small disc electrodes will be placed on the scalp.

DETAILED DESCRIPTION:
Objectives:

The purpose of this protocol is to improve understanding of the neurophysiological mechanisms that underlie the phenomenon of surround inhibition in the human motor cortex. It is known that patients with focal hand dystonia have abnormal motor surround inhibition. However, the physiology of this phenomenon still remains unclear. The 3 sub-studies proposed under this protocol will integrate several neurophysiological techniques to explore different aspects of motor surround inhibition. The objectives of sub-study 1 are (a) to identify the EEG correlate of motor SI (b) to determine the relationship between short interval intracortical inhibition (SICI) and SI, both of which are compromised in patients with FHD and (c) to determine if there is an oscillatory frequency band that is relevant for SI. The results from this sub-study will shed light on the inhibitory mechanisms that are critical for motor SI. Sub-study 2 is aimed at determining the influence of parietal conditioning on motor surround inhibition. If conditioning the parietal cortex enhances SI, we can conclude that the parieto-motor inhibitory network may be involved in motor SI and that this network could be affected in focal hand dystonia. Sub-study 3 will explore SI during different motor tasks.

Study population:

We intend to study up to 95 healthy volunteers in total. Up to 30 participants will be recruited for sub-study 1, 35 for sub-study 2, and 30 for sub-study 3.

Design:

Sub-study 1: This will be an exploratory study. Participants will perform an auditory cued index finger movement task and motor evoked potentials will be elicited by stimulating the motor hotspot of a surround muscle using transcranial magnetic stimulation (TMS). EEG will be recorded continuously. Single or paired TMS pulses (with postero-anterior or antero-posterior current) will be delivered either while the subject is at rest or at movement onset. TMS-evoked potentials (TEPs) will be obtained by time-locked averaging of all the trials in each condition. The amplitudes of the different peaks of the TEP will be compared across conditions which may be correlated with the degree of SI or SICI. The components of the TEP that are most relevant to motor SI will thus be identified.

Sub-study 2: This will be a hypothesis-driven study. Our primary hypothesis is that parietal conditioning will influence motor SI in healthy volunteers. Participants will perform an auditory cued index finger movement task and motor evoked potentials will be elicited by stimulating the motor hotspot of a surround muscle using transcranial magnetic stimulation. Two coils, one positioned over the motor cortex and the other over an inhibitory region of the inferior parietal lobule, will deliver TMS pulses at a fixed inter-stimulus interval. The pulses will be delivered either while the subject is at rest or at movement onset. The ratio of mean MEP amplitude obtained with parietal conditioning to that obtained with motor cortex stimulation alone at movement onset will reveal any parieto-motor influence on SI.

Sub-study 3: This will be an exploratory study. Participants will be asked to perform different motor tasks such as activating an intrinsic hand muscle at different levels of activation, sequential muscle activation or more complex tasks such as writing. Single TMS pulses will be delivered at primary motor cortex at rest, at the onset of the motor tasks or during the motor tasks. MEPs will be measured in the active and surround muscles. The ratios of MEP amplitudes during different levels of activation in the active and surround muscles will reveal

modulation of SI during these tasks.

Outcome measures:

For sub-study 1, our outcome measures will be (1) amplitudes of the different TEP peaks (2) degree of surround inhibition and short interval intracortical inhibition (3) correlation between them and relevant peak amplitudes (4) power and cortico-cortical coherence at different frequency bands.

MEP amplitude will be the primary outcome measure in sub-study 2 and 3.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age between 18 - 70 years.
* Right-handed (tested by the Edinburg handedness inventory).
* Able to give informed consent.
* Able to comply with all study procedures.
* Abstain from alcohol for at least 48 hrs prior to the study and caffeine on the day of the study (based on oral interview).

EXCLUSION CRITERIA:

* Illegal drug use within the past 6 months based on history alone. The intent is to exclude those with drug use that may affect study results.
* Self-reported consumption of >14 alcoholic drinks/week for a man and >7 alcoholic drinks/week for a woman.
* Abnormal findings on neurological examination.
* History of or current brain tumor, stroke, head trauma with loss of consciousness, epilepsy or seizures.
* Current episode of major depression or any major psychiatric illness.
* Taking medications that act directly on the central nervous system such as anti-epileptics, anti-histamines, anti-parkinsonian medication, muscle relaxants, medication for insomnia, anti-depressants, anti-anxiety medication.
* Presence of any metal in the eye or skull area such as a brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, metal fragments in the eye.
* Presence of pacemaker, intracardiac lines, implanted pumps or stimulators or metal objects inside the eye or skull.
* Known hearing loss.
* NIH employees and/or staff.
* Pregnancy

EXCLUSION CRITERIA for MRI (sub-study 2 only):

We will follow the Clinical Radiology/NMR Center guidelines for MR safety.

Some of the exclusions are:

* Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or metal fragments in the eye as these make having an MRI unsafe.
* Have metallic dental fillings which are likely to cause MRI artifacts
* Unable to lie flat on the back for the expected length of the experiment,
* up to 30 mins.
* Uncomfortable being in a small space for the expected length of the experiment, up to 30 mins.
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Substudy 2 TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal elicited by single /paired pulse TMS at rest or movement onset will give information about the corticospinal excitability. | throughout
  TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal elicited by single/paired pulse TMS at rest or movement onset will give information about the corticospinal excitability.
Substudy 1 EEG analysis: we will measure the latency and amplitude of the different components of the TMS-evoked potentials | throughout
  EEG: For the EEG analysis, we will measure the latency and amplitude of the different components of the TMS-evoked potentials. Time-frequency analysis on the collected EEG data will provide valuable information on which frequency bands are involved in the phenomenon of motor SI. The coherence calculated between relevant brain regions will also reveal information on the changes in cortical connectivity during the phenomenon of SI.
Substudy 1 TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal | throughout
  TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal elicited by single/paired pulse TMS will give information about the corticospinal excitability. The latency of the MEP will revealmore information on which neuronal networks were activated.
Substudy 3 TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal elicited by single pulse TMS at rest or during a motor task will give information about the corticospinal excitability. | throughout
  TMS: The amplitude of the motor evoked potential (MEP) in the EMG signal elicited by single pulse TMS at rest or during a motor task will give information about the corticospinal excitability.
Substudy 3 EMG: The EMG amplitude during certain tasks will reveal information about the level of muscle activation. | throughout
  EMG: The EMG amplitude during certain tasks will reveal information about the level of muscle activation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0031.html